CLINICAL TRIAL: NCT03773666
Title: A Feasibility Study of Durvalumab (MEDI4736) Alone or in Combination With Oleclumab (MEDI9447) as Neoadjuvant Therapy for Muscle-invasive Bladder Cancer (BLASST-2)
Brief Title: A Feasibility Study of Durvalumab +/- Oleclumab as Neoadjuvant Therapy for Muscle-invasive Bladder Cancer (BLASST-2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Xiao X. Wei, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-507
Record Dates: First submitted 2018-12-08; First posted 2018-12-12 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Muscle Invasive Bladder Cancer
Keywords: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Durvalumab (Experimental): -Durvalumab will be administered intravenously every 2 weeks, with 14 consecutive days defined as a treatment cycle
  Interventions: Drug: Durvalumab
- Durvalumab + Oleclumab (Experimental): * Durvalumab will be administered intravenously every 2 weeks, with 14 consecutive days defined as a treatment cycle
  * Oleclumab will be administered intravenously every 2 weeks, with 14 consecutive days defined as a treatment cycle
  Interventions: Drug: Durvalumab; Drug: Oleclumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab is a monoclonal antibody (an antibody is a protein produced by the body's immune system) that works by blocking the Programmed Cell Death Ligand 1 (PD-L1), a protein on cancer cells that stops the body's immune system from killing cancer cells.
  Other Names: MEDI4736
Drug: Oleclumab — Oleclumab is a monoclonal antibody that works by reducing the amount of adenosine, a small molecule called a metabolite that binds to adenosine receptors on immune cells to regulate the immune system and suppress the immune response. Reducing the amount of immunosuppressive adenosine can increase the body's immune response to kill cancer cells.
  Other Names: MEDI9447
  Arms: Durvalumab + Oleclumab

SUMMARY:
This research study is studying a new anti-cancer drug durvalumab (MEDI4736) with or without another new anti-cancer drug Oleclumab (MEDI9447) before surgery for bladder cancer.

The drugs involved in this study are:

* Durvalumab (MEDI4736)
* Oleclumab (MEDI9447)

DETAILED DESCRIPTION:
This research study is a Feasibility Study, which is the first time investigators are examining these drugs, Durvalumab (MEDI4736) and Oleclumab (MEDI9447) in patients with muscle-invasive bladder cancer (MIBC) cancer prior to surgery. Cisplatin-containing chemotherapy given before surgery is the standard of care in patients with MIBC because it increases the rate of cure after surgery. Participants may still be eligible for this study if their doctor determines that participants are able to receive cisplatin-containing chemotherapy, but the participants elect not to undergo chemotherapy before surgery, understanding the potential benefits of chemotherapy. The FDA (the U.S. Food and Drug Administration) has not approved Durvalumab (MEDI4736) for localized bladder cancer prior to surgery, but it has been approved for other uses, including for locally advanced or metastatic bladder cancer after progression on platinum-containing chemotherapy. The FDA (the U.S. Food and Drug Administration) has not approved Oleclumab (MEDI9447) as a treatment for any disease. Durvalumab is a monoclonal antibody (an antibody is a protein produced by the body's immune system) that works by blocking the Programmed Cell Death Ligand 1 (PD-L1), a protein on cancer cells that stops the body's immune system from killing cancer cells, to increase the body's immune response to prevent or slow down cancer growth. Oleclumab is a monoclonal antibody that works by reducing the amount of adenosine, a small molecule called a metabolite that binds to adenosine receptors on immune cells to regulate the immune system and suppress the immune response. Reducing the amount of immunosuppressive adenosine can increase the body's immune response to kill cancer cells. It is hoped that by combining Oleclumab with Durvalumab, an even greater immune response against the tumor will be generated. This research study is designed to see if the new anti-cancer drug Durvalumab (MEDI4736) with or without another new anti-cancer drug Oleclumab (MEDI9447) can be safely administered before surgery for bladder cancer

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in the study patients must fulfil all of the following criteria: Written informed consent and any locally-required authorization (e.g. HIPAA) obtained from the patient prior to performing any protocol-related procedures, including screening evaluations
* Age > 18 years at time of study entry
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (See Appendix A).
* Histologically confirmed bladder transitional cell carcinoma (TCC)

  ---Patients with mixed histology are required to have a component of TCC, and no component of small cell histology
* T2-T4a N0 M0 disease, considered appropriate and planned for radical cystectomy
* Ineligible for cisplatin-based chemotherapy, defined by any of the following:

  * Creatinine clearance (CL) <60 mL/min. GFR should be calculated from serum/plasma creatinine using the Cockcroft-gault formula.
  * CTCAE v5.0 Grade > 1 hearing loss
  * CTCAE v5.0 Grade > 1 neuropathy
  * NYHA Class > II cardiac dysfunction
* Patients not meeting the above criteria are eligible if she/he declines perioperative cisplatin-based chemotherapy after specific informed consent describing the known benefits of cisplatin-based chemotherapy.
* Adequate organ function laboratory values as defined below:

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count (ANC) 1.5 x (> 1500 per mm3)
  * Platelet count ≥100 x 109/L (>75,000 per mm3)
  * Albumin > 2.5 g/dL
  * International Normalized Ratio (INR) or activated partial thromboplastin time (aPTT) < 1.5 x ULN, unless the patient is receiving anticoagulation therapy provided INR or PTT is within the therapeutic range of the intended anticoagulant therapy.
  * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN)

    ---This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
  * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal
  * Measured creatinine CL >30 mL/min or Calculated creatinine CL>30 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

    * Males:
    * Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)
    * Females:
    * Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the postmenopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiationinduced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Availability of baseline archival tumor tissue obtained for correlative studies dated within 8 weeks of study registration.

  * Either FFPE tumor tissue block or a minimum of fifteen 5μm unstained FFPE slides and fifteen 10μm unstained FFPE slides with an associated pathology report is required.
  * Patients without adequate baseline tumor tissue or have archival tumor tissue >8 weeks from registration must undergo cystoscopic tumor biopsy, meeting the above tissue criteria.

Exclusion Criteria:

* Patients with primary TCC of the ureter, urethra, or renal pelvis without TCC of the bladder
* Inoperable tumor(s) with fixation to the pelvic wall on clinical exam
* Any previous systemic chemotherapy or radiotherapy for TCC of bladder
* Participation in another clinical study with an investigational product during the last 6 months
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease (e.g. cervical cancer in situ)
* Receipt of the last dose of intravesical chemotherapy or biologic therapy

  ≤ 42 days (6 weeks) prior to the first dose of study drug for patients who have received prior intravesical chemotherapy or biologic therapy (e.g. BCG)
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF)

  ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart) for durvalumab + oleclumab cohorts only. Patient safety and the cardiac EKG should be consulted as needed.
* Any unresolved toxicity NCI CTCAE version 5.0 Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  * Patients with Grade ≥2 neuropathy will be evaluated on a case-bycase basis after consultation with the Study Physician.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab and/or oleclumab may be included only after consultation with the Study Physician.
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g. hormone replacement therapy) is acceptable.
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogenic organ transplantation
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g. colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* History of leptomeningeal carcinomatosis
* Brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry.
* History of active primary immunodeficiency
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of study drug. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g. intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/ day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab

  + oleclumab or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
* Prior randomization or treatment in a previous durvalumab and/or oleclumab clinical study regardless of treatment arm assignment
* Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants Receiving at least One Dose of Study Therapy Followed by Surgery without Dose-Limiting Toxicity (DLT) up to Twelve Weeks Post-Radical Cystectomy (RC) | 2 years

SECONDARY OUTCOMES:
Number of Participants Receiving at least One Cycle of Study Therapy and Undergone RC Having <pT2N0 Disease at Time of RC | 2 years
Duration of Time of RC to Time of Documented Disease Relapse or Recurrence after RC | 2 years
Radiographic Progression by RECIST 1.1 Criteria from Time of Baseline Screening Imaging to the End of Treatment Imaging Pre-RC | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiao X Wei, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor-Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Requests may be directed to: [contact information for Sponsor-Investigator or designee].